CLINICAL TRIAL: NCT02354209
Title: Targeted Clinical Strategies and Low Abundance HIV Viraemia in Boosted-PI Therapy: an Observational Study
Brief Title: Targeted Clinical Strategies and Low Level Viraemia (LLV) in Boosted Protease Inhibitor Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SSAT 057
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-1 patients receiving bPI ARV: Non interventional study. Interventions will be clinically directed rather than by protocol.
  The following procedures will be carried out:
  1. Questionnaire on compliance and adherence
  2. Clinic Visit
  3. 20ml blood sample to be taken for Virological Resistance Testing and Next Generation Sequencing (only if plasma viral load is detectable)

SUMMARY:
The purpose of the study is to look at possible reasons why some HIV positive people who take their drugs properly and have no resistance to these drugs, still have low amounts of virus detectable in their blood. This is known as Low Level Viraemia (LLV). When low levels of HIV virus are present, some can mutate and make the drugs less effective (i.e. some variants of the virus become more resistant). Currently, however, these resistance mutations may be difficult to detect using standard tests for resistance because the amount of virus in the blood is very low and the standard tests aren't sensitive enough to pick up the mutations. The investigators will use more sensitive mutation detection methods, known as Next Generation Sequencing (NGS), to look at whether see if there are any low levels of drug resistant HIV virus developing in the blood when LLV occurs. The investigators will look at the different treatment strategies that are used in routine standard practice when LLV is detected and evaluate which is most effective in preventing development of resistance. The investigators hope this research will help to inform guidelines on the best way to treat HIV in the future.

DETAILED DESCRIPTION:
Phase of Study: Non-Drug Study

Objectives:

1. Primary To investigate the causes of low level viraemia (LLV) in HIV-infected individuals with no PI resistance associated mutations (RAMs) on conventional genotyping who have a detectable plasma HIV viral load (pVL) and report >95% adherence* to their ARV regimens containing a boosted protease inhibitor.

   *in case the questionnaire cannot be performed, clinical documentation of adherence will be used for interpretation of adherence level.
2. Secondary To observe the evolution in virologic and immunologic responses following routine clinical intervention in HIV-infected individuals with no primary protease inhibitor mutations (IAS, USA) on conventional genotyping who have a detectable plasma HIV viral load (pVL) and report >95% adherence* to antiretroviral regimens containing a boosted protease inhibitor.

   * in case the questionnaire cannot be performed, clinical documentation of adherence will be used for interpretation of adherence level.

Study Design: A multi-centre, non-drug, observational cohort study.

Methodology: HIV-infected individuals attending three selected HIV clinics at the Chelsea and Westminster Hospital, St Mary's Hospital and Guy's and St Thomas' Hospital over the duration of the study will be identified at weekly viral resistance meetings and routine clinic appointments if they demonstrate the following HIV pVL criteria:

1. An HIV pVL of 41-2000 copies/ml (c/ml) on two consecutive tests after being <40 c/ml on at least two occasions on a bPI-containing regimen
2. An HIV pVL of 41-2000 c/ml on two consecutive tests having never achieved <40 c/ml on a bPI-containing regimen after more than six months of treatment.

Eligible patients will be provided with a patient information sheet and a written consent form. Following consent:

1. Virologic and immunologic assessments will be collected from the clinical records available
2. Viral resistance test (VRT) (using VircoTYPE HIV-1 Virtual PhenotypeTM-LM for conventional genotyping and Ilumina MiSeq as next generation sequencing, NGS for minority species testing) will be performed on the first detectable HIV pVL(>40 c/mL) found in clinic and at 3 to 6 and 12 months later, if HIV pVL is still >40 c/mL.

Planned Sample Size: 120 to 240 samples over the one-year study period, with each centre providing 40 to 80 samples.

Summary of Eligibility Criteria: HIV-infected individuals with no primary protease inhibitor mutations (IAS, USA) on standard VRTs who have a detectable pVL and report >95% adherence* ARV regimens containing a boosted protease inhibitor with HIV VL criteria as detailed above. Individuals who have a detectable HIV VL after stopping ARV or having an 8-item Morisky score of above 2 (or <95% reported adherence will not be eligible.

*in case the questionnaire cannot be performed, clinical documentation of adherence will be used for interpretation of adherence level.

Number of Study Centres: Three

Duration of Study: One year from study approval. Samples for resistance testing will be collected over the duration of the study.

Criteria for Evaluation:

1. Emergence of new primary protease inhibitor mutations (IAS, USA) using NGS will be described.
2. Comparison of respective parameters (HIV VL and CD4 count) between different clinical interventions. The latter will not be dictated by the protocol but will be conducted as routine clinical practice.

Primary Endpoint:

Development of primary protease inhibitor mutations (IAS, USA) on NGS in HIV-infected patients with primary protease inhibitor mutations (IAS, USA) on standard VRTs who demonstrate LLV on ARV regimens containing a bPI.

Secondary Endpoints:

1. Proportion of patients achieving an undetectable HIV VL following an intervention during periods of LLV on ARV regimens containing a bPI
2. Evolution of CD4 cell count following an intervention during periods of LLV on ARV regimens containing a bPI.

Note: This is a non-drug study and no interventions will be dictated by this protocol.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in the study if ALL of the following criteria apply:

1. Chronic HIV-1 infection (adult male, female or transgender)
2. Age >18 years
3. Current HIV clinic attendee at the Chelsea and Westminster Hospital, St Mary's Hospital, and Guy's and St Thomas' Hospital [defined as at least 1 attended clinic visit since January 2010]
4. Receiving a boosted protease inhibitor-containing antiretroviral regimen (bPI ARV)
5. HIV plasma viral load (pVL) of 41-2000 copies/ml (c/ml) on two consecutive tests after being <40 c/ml on at least two occasions on a bPI-containing regimen OR HIV pVL of 41-2000 c/ml on two consecutive tests having never achieved <40 c/ml on a bPI containing regimen after more than six months of treatment.

Exclusion Criteria:

A subject will NOT be eligible for inclusion in this clinical trial if the following criteria apply:

1. Demonstrable detectable HIV VL after stopping ARV
2. 8-item Morisky score of 2 or more or documented poor adherence to combination ARV. (<95% adherence*)

   * in case the questionnaire cannot be performed, clinical documentation of adherence will be used for interpretation of adherence level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current HIV clinic attendee at the Chelsea and Westminster Hospital, St Mary's Hospital, and Guy's and St Thomas' Hospital [defined as at least 1 attended clinic visit since January 2010] receiving a boosted protease inhibitor-containing antiretroviral regimen (bPI ARV)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03-31 (Actual); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in primary protease inhibitor mutations on the HIV genome as defined by IAS-USA drug resistance mutations list. | Change between baseline and 12 months after first detectble viral load

SECONDARY OUTCOMES:
Proportion of patients achieving an undetectable HIV VL following an intervention following LLV on ARV regimens containing a bPI | 12 months after first detectable VL on bPI
Change in cell count following an intervention during periods of LLV on ARV regimens containing a bPI | Change in CD4 cell count from baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — Chelsea & Westminster Hospital
Locations (3):
- United Kingdom (3):
  - St Thomas Hospital, London
  - St Stephen's Centre, London
  - St Mary's Hospital, London